CLINICAL TRIAL: NCT07172347
Title: A Multicenter, Randomized, Double-blind, Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of VC005 Tablets in Subjects With Non-segmental Vitiligo
Brief Title: Efficacy and Safety Phase II Study of VC005 Tablets in Subjects With Non-segmental Vitiligo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-204
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Non-segmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VC005 Tablets Low Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets High Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets Placebo groups (Placebo Comparator)
  Interventions: Drug: VC005 Tablets Placebo

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 52 weeks
  Arms: VC005 Tablets High Dose groups; VC005 Tablets Low Dose groups
Drug: VC005 Tablets Placebo — VC005 Placebo groups repeat administration for 52 weeks
  Arms: VC005 Tablets Placebo groups

SUMMARY:
This clinical trial is a multicenter, randomized, double-blind, controlled phase II clinical study

ELIGIBILITY:
Inclusion Criteria:

* The subject understands and voluntarily signs the informed consent form (ICF) and is willing and able to comply with the study protocol.
* The subject is between 18 and 70 years of age (including borderline values) , regardless of gender.

Exclusion Criteria:

* Pregnant or lactating women, or subjects with pregnancy or lactation plans during the study period.
* All hair in the vitiligo area on the face is white.
* Those who are known or suspected to be allergic to the main ingredients and excipients of VC005 or similar drugs.
* Subjects who have previously received depigmentation treatment.
* Subjects who have received experimental drug administration or participated in device clinical trials within the first month or 5 half lives (whichever is longer) prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in facial vitiligo area score index (F-VASI) relative to baseline at week 24 | Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Peking University People's Hospital, Beijing, Beijng, China